CLINICAL TRIAL: NCT06011161
Title: The Brief Relationship Checkup: A 3-Session Program to Support Veteran Relationships
Brief Title: A Pilot of the Brief Relationship Checkup
Acronym: BRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canandaigua VA Medical Center (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dev J. Crasta, Principal Investigator, Canandaigua VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1469686
Record Dates: First submitted 2023-08-15; First posted 2023-08-25 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Relationship Distress
Keywords: Couple therapy; Primary Care

STUDY DESIGN:
Intervention Model Description: Single arm pilot. All participants will participate in the same treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brief Relationship Checkup (Experimental): Couples in the experimental condition will participate in three joint sessions of the Brief Relationship Checkup (BRC; Cordova 2014; Cigrang et al., 2016). This program has been tested in Air Force Primary Care but we do not know if veterans with mental health concerns will be able to attend it (feasibility), complete it safely (tolerability), and enjoy it (acceptability).
  Interventions: Behavioral: Brief Relationship Checkup (BRC)

INTERVENTIONS:
Behavioral: Brief Relationship Checkup (BRC) — The investigators are using the three 30-minute session protocol developed for Air Force Primary Care (Cigrang et al., 2016). Although it is simply referred to as the "Marriage Checkup" in that manuscript, the investigators use the name BRC to distinguish it from many other versions of Dr. James Cordova's Marriage Checkup (Cordova, 2014) adapted for different settings. Sessions in this version are briefer than other versions (30 mins vs. 60-90 mins) and this trial does not have any eligibility restrictions based on marital status.
  Other Names: Marriage Checkup; Relationship Checkup

SUMMARY:
The goal of this pilot trial is to study the Brief Relationship Checkup (BRC) program for Veterans with a combination of mental health and relationship concerns.

BRC has been studied in Air Force primary care, but has never been tested in the Department of Veterans Affairs. To prepare for a larger study of BRC, the investigators asked the following questions:

1. Can the research team deliver BRC to Veterans with mental health concerns? ("Feasibility")
2. What is the best way to measure BRC's impact? ("Pilot Outcomes")
3. Does BRC fit the needs of Veterans, and if not, what changes would fit participants' needs? ("Refinement")

Participants completed an initial interview, attended the BRC program, and completed a follow-up interview.

DETAILED DESCRIPTION:
PURPOSE: Relationship distress is a common problem for Veterans with mental health concerns. Relationship treatments like couple therapy are effective, but studies in the Department of Veterans Affairs (VA) find that they are infrequently used and have high dropout rates. One possible solution is for VA to offer Relationship Checkups, a short program that helps couples commit to concrete steps to improve their relationship. A brief version of the program designed for Air Force primary care -- called the Brief Relationship Checkup (BRC) for the purpose of the study -- may be an especially good fit for VA primary care or outpatient mental health teams.

RESEARCH PLAN: This study is a single-arm pilot trial of BRC in 20 couples. that are in distressed committed relationship where at least one partner is a Veteran who screens positive on a primary care mental health screen for common suicide risk factors including suicide ideation, depression, PTSD, or alcohol misuse (the "Identified Patient"). Participants provided initial ratings of outcomes in separate baseline sessions, completed BRC, and then completed separate post-treatment interviews and questionnaires.

SPECIFIC AIMS:

AIM 1: Evaluate feasibility of conducting a BRC trial in Veterans with mental health concerns. This includes recruitment rate, completion rate, and provider adherence to protocol.

AIM 2: Pilot outcomes that can be used to evaluate pre-post change in future studies of BRC. This includes relationship functioning, suicide risk factors, and treatment utilization.

AIM 3: Inform continued refinement of BRC to be suitable to the needs of Veterans and their partners. This includes examining current acceptability and using open-ended interviews.

ELIGIBILITY:
Inclusion Criteria:

1. BOTH PARTNERS must be age 18 or over
2. BOTH PARTNERS must demonstrate sufficient knowledge of English and cognitive capacity to understand the study through comprehension of consent questions
3. BOTH PARTNERS must self-identify as "in a committed relationship" with their partner for at least 6-months.
4. AT LEAST ONE PARTNER must report at least mild relationship distress on a satisfaction screen.
5. AT LEAST ONE PARTNER must have Veteran status
6. THE VETERAN PARTNER must screen positive on at least on a VA Primary Care Mental Health Screen (i.e., Patient Health Questionnaire(PHQ)-2 for Depression, PHQ Item 9 for Suicide Risk; Alcohol Use Disorders Identification Test Consumption Questions for At-Risk Drinking; or Primary Care-PTSD-5 for Potential PTSD)

Exclusion Criteria:

1. EITHER PARTNER reports that they are engaged in ongoing couple or family therapy.
2. EITHER PARTNER reports severe intimate partner violence in the last year.
3. EITHER PARTNER reports experiencing suicidal intent or suicidal attempts in the last month.
4. EITHER PARTNER experiences current psychosis.
5. EITHER PARTNER experiences current mania.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Finger Lakes Healthcare System (Canandaigua), Canandaigua, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
We will create deidentified datasets containing only variables used in a publication. This will be limited to the quantitative variables underlying publication to minimize likelihood of reidentification.
  Deidentified datasets will be stored in repositories if required for publication. Otherwise, they will be available on request to individual researchers with appropriate credentials.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data will be available beginning one year after publication.
Access Criteria: Researchers must demonstrate they are accessing the data for validation of results or other scientific/public purposes (e.g., replication of findings, incorporation of findings in meta-analyses).
  Data sets will not be shared prior to the facility Privacy Officer approval of the access request and deidentification steps.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: N/A. All participants are considered assigned to the treatment condition from the moment of couple enrollment.
Period: Overall Study
Arm/Group | Brief Relationship Checkup
Started | 40
Completed | 33
Not Completed | 7
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Population: This is a study of couples. Although all couples went through the same treatment, we provide separate demographics for Screened Veterans and Supporting Partners.
Groups:
- Screened Veteran: This is the first, VA-engaged Veteran partner of each couple that is referred to the study and has at least one positive VA mental health screen for depression, heavy drinking, PTSD, or relationship dissatisfaction. In the manuscript (Crasta et al., 2023), we refer to these participants as "VA-engaged Veterans," "Identified Patients," or "Patients" for short.
- Supporting Partner: This is the second partner that is referred to the study. This partner may or may not be a Veteran themselves. In the manuscript (Crasta et al., 2023), we refer to those participants as "Second Partners" or simply "Partners" for short.
- Total: Total of all reporting groups
Arm/Group | Screened Veteran | Supporting Partner | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.60 (13.68) | 41.45 (13.95) | 42.03 (13.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 17 | 20
  Male | 17 | 3 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 16 | 20 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 14 | 14 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Veteran Status [Count of Participants; unit: Participants]
  Veteran | 20 | 2 | 22
  Non-Veteran | 0 | 18 | 18

OUTCOME MEASURES:

1. Primary Outcome: Relationship Functioning
Description: Relationship Functioning will be measured using the Couples Satisfaction Index (CSI). The self-report scale has a minimum of 0 and a maximum of 161 with higher scores representing more satisfying relationships and scores < 104.5 classified as "distressed." The CSI is widely used in couple therapy research and is used routinely in VA care to evaluate Veterans' progress in evidence-based couple therapies.
Time Frame: Pre-treatment
Population: Full sample
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Second Partner: This is a romantic partner identified by the Screened Veteran to participate in the study with them and work on their relationship. This partner may or may not be a Veteran themselves. In the manuscript (Crasta et al., 2023), we also refer to these participants as "Supporting Partners" or simply "Partners" for short.
Arm/Group | Screened Veteran | Second Partner
Number analyzed (Participants) | 20 | 20
score on a scale | 84.99 (6.60) | 90.90 (6.60)

2. Primary Outcome: Relationship Functioning
Description: as for outcome 1
Time Frame: After Completing the BRC Program (1-3months after pre-treatment)
Population: Participants completing the measure at follow-up.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Screened Veteran | Second Partner
Number analyzed (Participants) | 15 | 16
score on a scale | 117.66 (6.97) | 106.81 (6.88)

3. Secondary Outcome: Emotional Intimacy/Mutual Responsiveness
Description: Emotional Intimacy will be measured using the Perceived Responsiveness & Insensitivity Scale (PRI). The PRI is an optimized measure of "Perceived Partner Responsiveness," a model of emotional intimacy that is widely used in the field to understand whether partners see one another as understanding/validating.
  The PRI has a minimum of 0 and a maximum of 80, with higher scores indicating greater sense of validation/understanding from one's partner.
Time Frame: Pre-treatment
Population: Whole sample
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Screened Veteran | Second Partner
Number analyzed (Participants) | 20 | 20
score on a scale | 41.64 (4.49) | 44.80 (4.49)

4. Secondary Outcome: Emotional Intimacy/Mutual Responsiveness
Description: Emotional Intimacy will be measured using the Perceived Responsiveness & Insensitivity Scale (PRI). The PRI is an optimized measure of "Perceived Partner Responsiveness," a model of emotional intimacy that is widely used in the field to understand whether partners see one another as understanding/validating.
  The PRI has a minimum of 0 and a maximum of 80, with higher scores indicating greater sense of validation/understanding (i.e., greater emotional intimacy).
Time Frame: After Completing the BRC Program (1-3months after pre-treatment)
Population: Participants completing the measure at follow-up.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Screened Veteran | Second Partner
Number analyzed (Participants) | 15 | 16
score on a scale | 58.87 (4.65) | 50.67 (4.61)

5. Secondary Outcome: Depressive Symptoms
Description: Depression will be measured using the 9-item Patient Health Questionnaire (PHQ-9). This self-report scale has a minimum of 0 and a maximum of 27 with higher scores representing greater number and frequency of depression symptoms and scores of 10 or higher representing moderate depression.
Time Frame: Pre-treatment
Population: Full sample
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Screened Veteran | Second Partner
Number analyzed (Participants) | 20 | 20
score on a scale | 11.00 (0.98) | 7.50 (0.98)

6. Secondary Outcome: Depressive Symptoms
Description: as for outcome 5
Time Frame: After Completing the BRC Program (1-3months after pre-treatment)
Population: Participants completing the measure at follow-up.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Screened Veteran | Second Partner
Number analyzed (Participants) | 15 | 16
score on a scale | 8.17 (1.08) | 4.24 (1.06)

7. Secondary Outcome: Perceived Burdensomeness
Description: Perceived burdensomeness will be measured with the burden-specific subscale of the Interpersonal Needs Questionnaire (INQ). This self-report scale has a minimum of 6 and a maximum of 42 with higher scores representing a stronger belief that one is a burden on others. Scores of 12 or higher predict a higher risk for developing suicidal ideation.
Time Frame: Pre-treatment
Population: All participants completing measure at baseline. Two participants missing data as measure is on last page.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Screened Veteran | Second Partner
Number analyzed (Participants) | 19 | 19
score on a scale | 11.14 (1.05) | 7.84 (1.07)

8. Secondary Outcome: Perceived Burdensomeness
Description: as for outcome 7
Time Frame: After Completing the BRC Program (1-3months after pre-treatment)
Population: All participants completing the measure at follow-up, with the exception of two screened Veterans who reported a 10-point reduction in burdensomeness who were removed from analysis in order to create a conservative estimate of reduction.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Screened Veteran | Second Partner
Number analyzed (Participants) | 13 | 16
score on a scale | 9.76 (1.09) | 7.06 (1.09)

9. Secondary Outcome: Thwarted Belongingness
Description: Thwarted belongingness will be measured with the belonging-specific subscale of the Interpersonal Needs Questionnaire (INQ). This self-report scale has a minimum of 9 and a maximum of 63 with higher scores representing a stronger feeling of loneliness and isolation. Scores of 36 or higher predict a higher risk for developing suicidal ideation.
Time Frame: Pre-treatment
Population: All participants completing measure at baseline. Two participants missing data as measure is on last page.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Screened Veteran | Second Partner
Number analyzed (Participants) | 19 | 19
score on a scale | 31.26 (2.43) | 28.32 (2.47)

10. Secondary Outcome: Thwarted Belongingness
Description: as for outcome 9
Time Frame: After Completing the BRC Program (1-3months after pre-treatment)
Population: Participants completing the measure at follow-up.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Screened Veteran | Second Partner
Number analyzed (Participants) | 15 | 16
score on a scale | 23.75 (2.55) | 23.50 (2.55)

11. Secondary Outcome: Suicide Ideation Severity
Description: Suicide ideation over the study will be monitored using the "Last Month" version of the Columbia Suicide Severity Rating Scale (CSSRS). This semi-structured interview has interviewers rate suicide ideation on a scale of 0 to 5, with scores of 3-5 placing individuals at high risk for attempt. VA hospitals use the C-SSRS across all clinics.
Time Frame: Pre-treatment
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Screened Veteran | Second Partner
Number analyzed (Participants) | 20 | 20
Participants
  No ideation (Score=0) | 18 | 20
  Passive Death Ideation (Score=1) | 1 | 0
  Ideation with Plan (Score=3) | 1 | 0

12. Secondary Outcome: Suicide Ideation Severity
Description: as for outcome 11
Time Frame: After Completing the BRC Program (1-3months after pre-treatment)
Population: Participants who completed as C-SSRS interview.
Measure: Count of Participants; unit: Participants
Arm/Group | Screened Veteran | Second Partner
Number analyzed (Participants) | 16 | 17
Participants
  No Ideation (Score=0) | 14 | 17
  Passive Death Ideation (Score=1) | 2 | 0
  Suicidal Ideation with Plan (Score=3) | 0 | 0

13. Secondary Outcome: Treatment Acceptability
Description: Treatment acceptability was assessed using the Client Satisfaction Questionnaire (CSQ, Larsen et al., 1979). Scores range from 1-4 with scores greater than 3 representing satisfaction with the treatment.
Time Frame: After Completing the BRC Program (1-3months after pre-treatment)
Population: All participants completing the follow-up survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Screened Veteran | Second Partner
Number analyzed (Participants) | 15 | 16
score on a scale | 3.49 (0.50) | 3.43 (0.52)

14. Other Pre Specified Outcome: Number of Mental Health and Family Contacts
Description: Treatment engagement in mental health services will be assessed through a review of the electronic medical record. Staff will review appointments (e.g., individual, group, assessments) with a specific focus on general mental health services and couple/family support services (including Caregiver Support program and Intimate Partner Violence Assistance Program).
Time Frame: 90 day period before pre-treatment session
Population: Participants who completed treatment and had accessible charts in the VA medical record
Measure: Mean (Standard Deviation); unit: days of care
Arm/Group | Screened Veteran | Second Partner
Number analyzed (Participants) | 18 | 3
days of care | 3.39 (3.11) | 0.33 (0.58)

15. Other Pre Specified Outcome: Number of Mental Health and Family Contacts
Description: as for outcome 14
Time Frame: 90 day period after final treatment session (earliest window 1-4mo after pre-treatment session and latest window 3-6mo)
Population: Participants who completed treatment and had accessible charts in the VA medical record
Measure: Mean (Standard Deviation); unit: days of care
Arm/Group | Screened Veteran | Second Partner
Number analyzed (Participants) | 18 | 3
days of care | 4.78 (4.33) | 2.67 (3.79)

ADVERSE EVENTS:
Time Frame: Study duration from first to last assessment (1-3 months).
Description: In addition to non-systematic assessment of adverse events broadly used by the (i.e., untoward or unfavorable medical occurrence in a participant), we also used systematic assessments to monitor for any intimate partner violence, self-harm, or suicidal behavior from first visit to last visit.
Arm/Group | Screened Veteran | Second Partner
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Screened Veteran (N=20) | Second Partner (N=20)
Intimate Partner Violence Event (Social circumstances) | 1 (1) | 1 (1) — Occurrence of physical conflict behavior even if it does not lead to medical complications. Our single violence event is marked as a negative event for both partners in the couple.
Non-Suicidal Self-Injury (Psychiatric disorders) | 0 (0) | 0 (0) — Any form of intentional self-injury without suicidal intent, even if it does not lead to medical consequences or hospitalization.
Suicidal Behavior (Psychiatric disorders) | 0 (0) | 0 (0) — Any suicidal attempt, self/other interrupted attempt, or preparatory behavior even if it does not result in hospitalization or medical consequences .

LIMITATIONS AND CAVEATS:
This study is a small pilot without a comparison group and half of the Screened Veterans were participating in individual therapy. Therefore, it is possible that some of these couples may have been expected to naturally improve over time, and it is unclear how much of the improvements seen in this ClinicalTrials.gov registration are due to the treatment itself.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT06011161/Prot_SAP_001.pdf
  • Informed Consent Form (2020-03-27): https://cdn.clinicaltrials.gov/large-docs/61/NCT06011161/ICF_000.pdf